CLINICAL TRIAL: NCT06637891
Title: The Effect of Mandala Coloring on Postpartum Blues: a Randomized Controlled Trial
Brief Title: Mandala Coloring and Postpartum Blues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Ayca Solt Kirca, Asssociate professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KırklareliAS-14
Record Dates: First submitted 2024-10-05; First posted 2024-10-15 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Post Partum Depression; Depression, Anxiety
Keywords: Mandala coloring; postpartum blues
MeSH Terms: conditions — Depression, Postpartum; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala coloring group (Experimental): Mandala painting will be applied to postpartum women who have postpartum blues
  Interventions: Other: Mandala coloring
- Control group (No Intervention): Participants in this group will consist of people who do not routinely do any practice on their own to reduce postpartum blues symptoms.

INTERVENTIONS:
Other: Mandala coloring — Participants will be asked to choose the pages they want from 12 colored felt-tip pen paint sets and 16 mandala coloring pages given to each participant by the researcher for 2 weeks, 3 days a week, at any time of the day and for an average of 20-30 minutes each time, and paint them in the colors they want.
  Arms: Mandala coloring group

SUMMARY:
One of the art therapy techniques that can provide psychological support and healing is mandala painting. Mandala is a Sanskrit word meaning 'circle'. The purpose of the circle is to encourage meditation, concentration and integration by narrowing or limiting the visual field towards the centre. In mandala painting, the individual can focus on the lines, stay in the moment, separate themselves from the concerns of the past and future and allow them to recall the consciousness of the moment. Studies in the literature have reported that making mandalas is an effective method for reducing negative mood and anxiety in people.This study was planned as a randomized controlled study to help women who experience postpartum sadness get through this period more easily.

DETAILED DESCRIPTION:
One of the art therapy techniques that can provide psychological support and healing is mandala painting. Mandala is a Sanskrit word meaning 'circle'. The purpose of the circle is to encourage meditation, concentration and integration by narrowing or limiting the visual field towards the center. In mandala painting, the individual can focus their attention on the lines, stay in the moment, separate themselves from the concerns of the past and future and ensure that they remember the consciousness of the moment again. The energy and emotions of the individual can change with the rich variety of colors used in mandala painting. It can help the individual achieve spiritual calmness by silencing the chaos and sounds that disturb them. Studies in the literature have reported that mandala painting is an effective method in reducing negative moods and anxiety in individuals. Gray-Foti found in his study that mandala painting reduced the anxiety levels of new mothers and increased their self-confidence, while Özsavran and Akyıldız found that it increased the comfort and resilience of mothers with special needs children. In a meta-analysis study evaluating the effect of mandala painting on state anxiety in adults, it was determined that it was effective in reducing anxiety. However, no study has been found investigating the effect of mandala coloring on postpartum sadness.This study was planned as a randomized controlled study to help women who experience postpartum sadness get through this period more easily.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35,
* Being between the 1st and 14th days postpartum
* Being able to read, understand and write Turkish,
* Having given birth at term (single birth at 38 weeks and above),
* Having given birth by normal vaginal delivery or cesarean section after an uncomplicated pregnancy
* Scoring 13 points or above on the Edinburgh Postpartum Depression Scale
* Scoring 3 points or above on the Stein Blues Scale
* Having stable vital signs, not having undergone infertility treatment, not having a chronic disease (such as hypertension, diabetes), not experiencing severe depression, anxiety and stress, not having any chronic disease or not having a disease that may cause cognitive impairment (such as delirium, dementia, mental retardation), not having serious complications in the mother and volunteering to participate in the study will be included in the study.

Exclusion Criteria:

* Not meeting inclusion criteria

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 77 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Introductory Information form A form that includes questions about women's socio-demographic and pregnancy and characteristics. Introductory Information form | between 1 to 4 weeks
  A form that includes questions about women's socio-demographic and pregnancy and characteristics. The survey consists of questions covering the personal characteristics, obstetric characteristics and psycho-social characteristics of new mothers.
Stein Blues Scale | between 1 to 4 weeks
  The scale consists of two sections with a total of 13 questions. The first eight questions are Likert-type questions that examine mood symptoms. The second section investigates the presence of symptoms of headache, restlessness, difficulty in concentration, forgetfulness and confusion with five questions answered with yes/no. The scoring of the section with Likert-type questions varies between 0 and 4, and if there are symptoms in the last five questions, 1 point is added to the total score for each. The minimum score is 0, and the maximum score is 26. Patients are asked to answer the scale thinking only about that day.
Edinburgh Postpartum Depression Scale | between 1 to 4 weeks
  Responses to the 4-point Likert-type scale consisting of ten questions are scored between 0 and 3. The cut-off score for the scale is taken as 12/13. If the score is 12 and below, the patient is not considered at risk for postpartum depression, and if it is 13 and above, the patient is considered at risk for postpartum depression. Scores from 0 to 30 are taken from the scale.

CONTACTS AND LOCATIONS:
Overall Officials: ELIF DAGLI, P, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No